CLINICAL TRIAL: NCT05189210
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Prospective, 52-Week, Phase 2 Clinical Study to Evaluate the Safety and Efficacy of GV1001 Administered Subcutaneously for the Treatment of Mild to Moderate AD
Brief Title: GV1001 Subcutaneous(SC) for the Treatment of Mild to Moderate Alzheimer's Disease (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GemVax & Kael (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GV1001-AD-CL2-007
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Mild to Moderate Alzheimer's Disease
Keywords: Alzheimer's Disease; GV1001
MeSH Terms: conditions — Alzheimer Disease | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo SC injection administered once weekly for 4 weeks then every 2 weeks through Week 50
  Interventions: Drug: GV1001 Placebo
- GV1001 0.56 mg (Experimental): GV1001 0.56 mg SC injection administered once weekly for 4 weeks then every 2 weeks through Week 50
  Interventions: Drug: GV1001 0.56mg
- GV1001 1.12 mg (Experimental): GV1001 1.12 mg SC injection administered once weekly for 4 weeks then every 2 weeks through Week 50
  Interventions: Drug: GV1001 1.12mg

INTERVENTIONS:
Drug: GV1001 Placebo — 0.9% normal saline
  Other Names: Normal saline
  Arms: Placebo
Drug: GV1001 0.56mg — Lyophilized peptide from hTERT
  Other Names: Tertomotide 0.84mg
  Arms: GV1001 0.56 mg
Drug: GV1001 1.12mg — Lyophilized peptide from hTERT
  Other Names: Tertomotide 1.68mg
  Arms: GV1001 1.12 mg

SUMMARY:
The current study is being conducted by the Sponsor to evaluate the efficacy and safety of GV1001 (0.56 mg and 1.12 mg) administered subcutaneously as a treatment for mild to moderate Alzheimer's disease (AD). Studies using in vivo and in vitro AD models have shown that GV1001 inhibits neurotoxicity, apoptosis, and the production of reactive oxygen species induced by amyloid beta (Aβ) in neural stem cells by mimicking the extra-telomeric functions of human telomerase reverse transcriptase (hTERT). In nonclinical studies, using both mild (early stage) and severe (late stage) AD mouse models, GV1001 was shown to improve cognitive function and memory, as well as significantly reduce the amount of Aβ and tau proteins. The multifunctional effect of GV1001 makes it a promising therapeutic option for the treatment for AD. In a completed Phase 2 study conducted in Korea, GV1001 showed significant improvement in change from baseline of Severe Impairment Battery score at Week 24 and demonstrated a clinically acceptable safety profile in patients with moderate to severe AD.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group Phase 2 study in participants with mild to moderate AD. The study will consist of a screening visit (up to 60 days prior to first dose), a 52-week double-blind treatment period, and an end-of-study (EOS) visit 2 weeks after the last dose of study drug. Eligible participants will be randomized in a 1:1:1 ratio to receive GV1001 0.56 mg, GV1001 1.12 mg, or placebo (normal saline) every week for 4 weeks beginning on Day 1 (of Week 1) followed by every 2 weeks through Week 50.

Prior to randomization, eligibility of potential participants will be confirmed through an adjudication process in which screening data (eg, MMSE, magnetic resonance imaging [MRI] scans, positron emission tomography [PET] scans) obtained to evaluate AD status are reviewed by a medical monitor. The medical monitor will review the subject eligibility form completed by the Investigator prior to randomization and provide an independent assessment of the participant's eligibility and may request exclusion of a participant from entry into the study. A central independent reader will review MRI to confirm eligibility. Investigators must not randomize a participant prior to receipt of this independent confirmation of the participant's eligibility. Results from MRI, Aβ positron emission tomography (PET) scan, cerebrospinal fluid (CSF) examination or genetic testings performed within the 2 years prior to screening will also be used to confirm eligibility. If no historical results are available, participants will undergo a MRI or an Aβ PET scan at screening.

If a participant discontinues treatment prematurely, the participant will be asked to continue with the scheduled study visits until the EOS visit. If a participant discontinues the study prematurely (except for those who withdraw their consent), the participant will be asked to come for an early termination (ET) visit for efficacy scale and safety assessments. These assessments are the same as those scheduled at the primary endpoint (PE) visit at Week 52. If the ET visit takes place within 4 weeks after a completed protocol scheduled visit with efficacy assessments, efficacy scale assessments are not required at the ET visit.

For an individual participant, the maximum duration of study participation is approximately 14.5 months, including an up to 60-day screening period.

An independent Data and Safety Monitoring Board (DSMB) review to evaluate safety data will be performed when at least 90 participants (50%) have either completed Week 26 or have discontinued the study. The DSMB may recommend early stopping of the study for safety reasons.

Efficacy evaluations will be performed at baseline, Week 12, Week 26, Week 38, and Week 52 using the cognitive subscale of the Alzheimer's Disease Assessment Scale [ADAS-cog11]), assessment of activities of daily living (ie, Amsterdam Instrumental Activities of Daily Living Questionnaire [A-IADL-Q]), and global ratings of dementia (ie, Clinical Dementia Rating-Sum of Boxes [CDR-SB], Neuropsychiatric Inventory [NPI], Mini-Mental State Examination [MMSE], Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change/Clinician's Interview-Based Impression of Change - Plus Family Input [ADCS-CGIC/CIBIC-Plus], and Quality of Life in Alzheimer's Disease [QoL-AD]). The ADAS-cog11 scale will be evaluated by a central independent reader for each visit. At the visits where several efficacy assessments are administered, every effort should be made to perform the efficacy evaluations in the same order at each visit (ADAS-cog11, A-IADL-Q, NPI, MMSE, CDR-SB, ADCS-CGIC/CIBIC-Plus, and QoL-AD).

Safety will be assessed throughout the study by monitoring for AEs, laboratory evaluations, electrocardiogram (ECG) findings, and vital signs measurements. Suicidal ideation and behavior will be assessed using the C-SSRS. Blood and CSF samples will be collected to evaluate the effect of GV1001 on analysis of biomarkers of AD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 55 to 85 years of age (both inclusive) at the time of signing the informed consent.
2. Diagnosis of probable AD based on NINCDS-ADRDA criteria (a and b) as determined by a neurologist, geriatrician, psychiatrist, or clinician approved by the Sponsor or designee.

   a. Presence of an early and significant episodic memory impairment that includes the following features: i. Gradual and progressive change in memory function reported by patients or informants over >6months.

   ii. Objective evidence of significantly impaired episodic memory on testing: this generally consists of recall deficit that does not improve significantly or does not normalize with cueing or recognition testing and after effective encoding of information has been previously controlled.

   iii. The episodic memory impairment can be isolated or associated with other cognitive changes at the onset of AD or as AD advances.

   b. One or more findings for probable AD by either MRI, Aβ PET scan, historical CSF results, or a historical genetic test in the 2 years before screening, or an MRI or Aβ PET scan at screening. The MRI must have findings consistent with AD and without any other disease that may cause dementia. The Aβ PET scan and historical CSF results must be consistent with the presence of amyloid pathology.
3. Mild or moderate dementia as evidenced by MMSE score ≥13 to ≤24 at screening (Visit 1).
4. Not applicable.
5. Not applicable.
6. If receiving an approved medication for AD (ie, donepezil, galantamine, rivastigmine, memantine, or memantine/donepezil combination product), must be on the medication with a stable dose for at least 12 weeks before the screening visit (dosing should remain stable throughout the study).
7. If receiving an OTC supplement for cognition (eg, gingko biloba, omega-3 polyunsaturated fatty acid, vitamin E, curcumin), must not be exceeding the recommended dose for at least 12 weeks prior to screening visit.
8. Able to visit the study center and undergo cognitive, functional, and other tests specified in the protocol.
9. Has a caregiver who:

   * Agrees to accompany the participant to all study visits and able to supervise the participant's compliance with the study procedures and provide detailed information about the participant.
   * Either lives with the participant or sees the participant on average for ≥1 hour/day ≥3 days/week, or in the Investigator's opinion, the extent of contact is sufficient to provide meaningful assessment of changes in participant behavior and function over time and provide information on safety and tolerability.
   * Is able to read, understand, and speak the designated language at the study center.
   * Caregiver must be cognitively able to fulfill the requirements of the study.
10. A male participant must agree to use a highly effective contraception method as detailed in Appendix 3 during the treatment period and for at least 3 months after the last dose of study treatment and refrain from donating sperm during this period.
11. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    * Not a woman of childbearing potential as defined in Protocol Appendix 3. OR
    * A WOCBP who agrees to use a highly effective contraception method as detailed in Appendix 3 during the treatment period and for at least 3 months after the last dose of study treatment.
12. A WOCBP must have a negative serum pregnancy test (beta-human chorionic gonadotropin [β-hCG]) at screening (Visit 1) and a negative urine pregnancy test at Visit 2 before randomization, and must use medically accepted means of contraception throughout the study.
13. Written informed consent provided by participant (or legal representative) and caregiver prior to any study-specific procedures.
14. Participants in France must belong to a social security scheme.

Exclusion Criteria:

1. Any other cause of dementia shown by MRI/CT findings within 2 years of screening and neurological examination at screening and Day 1.

   * Possible, probable, or definite vascular dementia according to the National Institute of Neurological Disorders and Stroke and Association Internationale pour la Recherché et l'Enseignement en Neurosciences (NINDS-AIREN) criteria.
   * Evidence of significant abnormality that would suggest another potential etiology for dementia (eg, evidence of cerebral contusion, encephalomalacia, aneurysm, vascular malformation, >5 microhemorrhages, macrohemorrhage, single infarct >1 cm3).
   * Other central nervous system diseases that may cause cognitive impairment (eg, cerebrovascular disease including cerebrovascular dementia, Parkinsonism, Huntington's disease, subdural hematoma, normal pressure hydrocephalus, brain tumor, Creutzfeldt-Jakob disease).
2. Concurrent or history of schizophrenia or bipolar disorder; OR any other clinically significant psychiatric conditions that in the Investigator's opinion prevents the participant from participating, or is likely to confound interpretation of drug effect or affect cognitive assessments or participant safety; OR the presence or history of suicidal attempts or suicidal ideation evidenced by endorsing Items 4 or 5 of the C-SSRS at screening or Day 1, endorsing any suicidal behavior item on the C-SSRS Since Last Visit form on Day 1, or any suicide attempt within 2 years prior to screening.
3. Vitamin B12, folic acid, syphilis serology, and thyroid stimulating hormone (TSH) results that are thought to contribute to the severity of dementia or cause dementia. Participants may be enrolled if in the Investigator's medical judgment, the abnormal laboratory values are not the cause of the cognitive symptoms.
4. History of known or suspected seizures including febrile seizures (excluding self-limited childhood febrile seizures), a history of significant head trauma with loss of consciousness or recent unconsciousness that is not explained.
5. Acute or unstable cardiovascular disease, active peptic ulcer, uncontrolled hypertension, uncontrolled diabetes or insulin dependent patients or any medical condition that may interfere with the completion of the clinical study.
6. Known allergies, hypersensitivity, or intolerance to GV1001 or similar products or excipients.
7. History of alcohol, substance abuse or dependence as per DSM-V criteria (except nicotine dependence) within the last 2 years.
8. Concurrent malignancies or invasive cancers diagnosed within the past 5 years except for non-metastatic basal cell carcinoma or squamous cell carcinoma of skin, in situ carcinoma of the uterine cervix or non-metastatic prostate cancer.
9. Sexually-active WOCBP or man capable of fathering a child who do not consent to using medicinally acceptable contraception (such as surgical sterilization, intrauterine contraceptive device, condom or diaphragm, an injectable or inserted contraceptive) during the study and for 3 months after the last dose of study treatment.
10. Pregnant, breast feeding, or planning a pregnancy or fathering a child while enrolled in the study or for 3 months after the last dose of study treatment.
11. Use of anxiolytics, narcotics, or sleep aids in a manner that would interfere with cognitive testing, in the opinion of the Investigator. Atypical antipsychotics may be used at the discretion of the Investigator. Tricyclic antidepressants and monoamine oxidase (MAO) inhibitors are prohibited
12. Previous treatment with GV1001.
13. Received an investigational product for AD within the last 6 months.
14. Participated in another clinical study within 4 weeks prior to this study.
15. Treated with aducanumab or participated in a clinical study with aducanumab.
16. Renal impairment (creatinine clearance [CrCL] <30 mL/min).
17. Severe liver dysfunction (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >2 times the upper limit of normal [ULN]).
18. Body weight ≤35 kg.
19. Resides in a moderate to high dependency continuous care facility (residence in low grade assisted living facility where there is sufficient autonomy to permit valid evaluation of activities of daily living is allowed).
20. Any other reason that in the opinion of the Investigator would make the participant ineligible to participate or to complete this study.

    [Additional Exclusion Criterion for Sites in France]
21. Patients deprived of their liberty by a judicial or administrative decision, and/or persons under psychiatric care within the meaning of Article L1121-6 of the Public Health Code.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ADAS-Cog11 score at Week 52 | Baseline, Week 12, Week 26, Week 38, and Week 52
  The Alzheimer's Disease Assessment Scale (ADAS) consists of 2 parts, a cognitive subscale and a behavioral subscale. The 11-item cognitive subscale (ADAS-cog) of the ADAS instrument will be used in this study. The ADAS-cog11 is a widely accepted performance-based assessment of cognition used in clinical studies for the treatment of participants with AD.
  The ADAS-cog11 (score range) consists of word recall (0-10) and word recognition memory tests (0-12), object and finger naming (0-5), commands (0-5), constructional praxis (0-5), ideational praxis (0-5), orientation (0-8), remembering test instructions (0-5), spoken language ability (0-5), comprehension of spoken language (0-5) and word finding difficulty (0-5). The maximum possible total score is 70, with a higher ADAS-cog11 score indicating worse cognitive function.

SECONDARY OUTCOMES:
Change from baseline in A-IADL-Q score at Week 12, Week 26, Week 38, and Week 52 | Baseline, Week 12, Week 26, Week 38, and Week 52
  Assessment of cognitively complex "instrumental activities of daily living" (IADLs), such as managing personal finances, using mobile phones, or even doing grocery shopping, is related to quality of life, caregiver burden, and resource utilization and is a relevant area to assess in AD clinical trials. There are various well validated IADL scales, but some are outdated as they do not assess current daily tasks.
  The Amsterdam IADL Questionnaire (A-IADL-Q) is an adaptive and computerized questionnaire designed to assess impairments IADL in patients with cognitive decline due to mild dementia. The questionnaire is completed by a caregiver and consists of 70 items in 7 categories (time needed 20-25 minutes).
Change from baseline in CDR-SB score at Week 12, Week 26, Week 38, and Week 52 | Baseline, Week 12, Week 26, Week 38, and Week 52
  The Clinical Dementia Rating (CDR) is a 5-point global rating scale used to characterize 6 domains of cognitive and functional performance applicable to AD and related dementias: memory, orientation, judgment & problem solving, community affairs, home & hobbies, and personal care. The information needed to make each rating is obtained through a semi-structured interview of the participant and a reliable informant or collateral source (eg, family member). The CDR rater should be trained to administer the semi-structured interview and should be blinded to results of other assessments.
  For each domain, a rating is assigned to quantify the severity of impairment/dementia (0=no impairment; 0.5=very mild impairment; 1=mild impairment; 2=moderate impairment; and 3=severe impairment). The sum of the ratings for the 6 domains is the Clinical Dementia Rating-Sum of Boxes (CDR-SB) score.
Clinical worsening, defined as ≥4 points change from baseline in the ADAS-cog11 score at Week 12, Week 26, Week 38, and Week 52 | Baseline, Week 12, Week 26, Week 38, and Week 52
  The Alzheimer's Disease Assessment Scale (ADAS) consists of 2 parts, a cognitive subscale and a behavioral subscale. The 11-item cognitive subscale (ADAS-cog) of the ADAS instrument will be used in this study. The ADAS-cog11 is a widely accepted performance-based assessment of cognition used in clinical studies for the treatment of participants with AD.
  The ADAS-cog11 (score range) consists of word recall (0-10) and word recognition memory tests (0-12), object and finger naming (0-5), commands (0-5), constructional praxis (0-5), ideational praxis (0-5), orientation (0-8), remembering test instructions (0-5), spoken language ability (0-5), comprehension of spoken language (0-5) and word finding difficulty (0-5). The maximum possible total score is 70, with a higher ADAS-cog11 score indicating worse cognitive function.
Change from baseline in NPI score at Week 12, Week 26, Week 38, and Week 52 | Baseline, Week 12, Week 26, Week 38, and Week 52
  The NPI is a validated informant-based interview that assesses behavioral symptoms of dementia. It covers 12 domains.
  The NPI is administered to the participant's caregiver and includes an integrated caregiver distress measure. For each domain, abnormal behavior is noted to be absent (score=0) or present. If present, the frequency (rarely=1, sometimes=2, often=3, and very often=4), severity (mild=1, moderate=2, and severe=3), and associated caregiver distress (0=not at all, 1=minimally, 2=mildly, 3=moderately, 4=severely, and 5=very severely or extremely) are to be rated.
  The product of frequency and severity (maxi.=12) is calculated for each domain. A total NPI was the sum of the frequency and severity products (maxi. =144). A higher NPI score indicates a greater degree of behavioral disturbances.
Change from baseline in MMSE score at Week 12, Week 26, Week 38, and Week 52 | Baseline, Week 12, Week 26, Week 38, and Week 52
  The MMSE is a brief test of cognitive function, defined as the sum of 11 items: orientation in time and place, registration, attention and concentration, recall, naming 2 objects, repetition, 3-stage command, reading, writing and copying. Scores range from 0 to 30; higher scores indicate better cognitive function.
Change from baseline in ADCS-CGIC/CIBIC-Plus score at Week 12, Week 26, Week 38, and Week 52 | Baseline, Week 12, Week 26, Week 38, and Week 52
  The CIBIC-Plus is used as a measure of global clinical status. It is an independent, semi-structured medical interview that is used to assess changes in the participant's condition during a clinical study. An independent, experienced, and properly trained rater will provide a global impression of the participant's condition based on separate interviews with the participant and caregiver.
  The rater is not to elicit caregiver's opinion of the participant's condition but only factual information about the study participant's functioning.
  The change from baseline in CIBIC-Plus is rated on a 7-point scale: 1=markedly improved, 2=moderately improved, 3 = minimally improved, 4=no change, 5=minimally worse, 6=moderately worse, and 7=markedly worse.
Change from baseline in QoL-AD score at Week 26 and Week 52 | Baseline, Week 26, and Week 52
  The QoL-AD includes the participant's and caregiver's appraisal of the participant's physical condition, mood, interpersonal relationships, ability to participate in meaningful activities, financial situation, and an overall assessment of self as a whole and life quality as a whole. It seems to be reliable and valid for individuals with MMSE scores greater than 10. The measure has 13 items, rated on a 4-point scale (poor, fair, good, excellent), with "l" being poor and "4" being excellent. Total scores range from 13 to 52. Separate scores are calculated for participant and caregiver reports.

CONTACTS AND LOCATIONS:
Overall Officials: Jeongmi Kim, Study Director — GemVax & KAEL Co., Ltd.
Locations (35):
- United States (12):
  - First Choice Neurology - Aventura Neurologic Associates, Adventura, Florida
  - Finlay Medical Research Corporation - Greenacres, Greenacres City, Florida
  - Outpatient Psy Care, Miami, Florida
  - Finlay Medical Research Corporation - Miami Dade, Miami, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Neurostudies - Port Charlotte, Port Charlotte, Florida
  - Palm Beach Neurology and Premiere Research Institute, West Palm Beach, Florida
  - Accel Research Sites (ARS) - NeuroStudies, Decatur, Georgia
  - Global Medical Institutes - Princeton Medical Institute, Princeton, New Jersey
  - Flourish Research - Alzheimer's Memory Center/AMC Research, LLC, Charlotte, North Carolina
  - Neurology Clinic - Cordova, Cordova, Tennessee
- Terveystalo Oulu, Oulu, Finland
- France (2):
  - Hôpital La Grave, Toulouse, Midi-Pyrenees
  - Hôpital Pierre Wertheimer, Bron, Rhône
- Casa di Cura iGEA SpA c/o Casa di Cura Privata del Policlinico, Milan, Italy
- Netherlands (3):
  - Brain Research Center - Amsterdam, Amsterdam, North Holland
  - Brain Research Center - Zwolle, Zwolle, Overijssel
  - Brain Research Centre - Den Bosch, Amsterdam
- Poland (6):
  - Centrum Medyczne Neuromed - Ośrodek Badań Klinicznych, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Wroctawskie Centrum Alzheimerowskie (WCA), Wroclaw, Lower Silesian Voivodeship
  - Galen Clinic, Lublin, Lublin Voivodeship
  - Centrum Medyczne Neuroprotect, Warsaw, Masovian Voivodeship
  - Niepubliczny Zakład Opieki Zdrowotnej NOVO-MED, Katowice, Silesian Voivodeship
  - Clinhouse Centrum Medyczne, Zabrze, Silesian Voivodeship
- Portugal (3):
  - Unidade Local de Saúde de Santa Maria, E. P. E. - Hospital de Santa Maria, Lisbon, Lisbon District
  - Hospital Pedro Hispano, Senhora da Hora, Porto District
  - Unidade Local de Saúde de Braga, E. P. E (Hospital de Braga), Braga
- Spain (7):
  - Hospital Universitario Quirónsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Fundacio ACE, Barcelona
  - Hospital Victoria Eugenia, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No